CLINICAL TRIAL: NCT04364672
Title: Molecular Neuroimaging to Assess the Link Between Neuroinflammation and Cognitive Impairment in Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of recruitment and funding
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R20-003
Record Dates: First submitted 2020-03-02; First posted 2020-04-28 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women with stage 1-4 newly diagnosed breast cancer (Experimental)
  Interventions: Drug: 18F-labeled DPA-714 PET scan

INTERVENTIONS:
Drug: 18F-labeled DPA-714 PET scan — One PET with [18F]DPA-714 before chemotherapy treatment begins. One more PET with [18F]DPA-714 within 4 weeks after completing NACT including at least 2 cycles administered; before surgery

SUMMARY:
This clinical study will use the small molecule translocator protein (TSPO) ligand, 18F-labeled DPA-714, to visualize and quantify neuroinflammation in treatment naive women with stage II-III newly diagnosed breast cancer (without brain metastases) prior to starting neoadjuvant chemotherapy treatment (baseline) and within 4 weeks after finishing neoadjuvant chemotherapy (NACT) with at least 2 cycles administered and before surgery. . The TSPO PET and MRI data acquired through this study will be correlated with cognitive test data, clinical data, and genetic testing collected in this study. We will enroll 20 participants in this study (20 participants with breast cancer).

Study Aim 1:

To examine the association between neuroinflammation and cancer related cognitive impairment (CRCI) in women with breast cancer before and after undergoing chemotherapy treatment.

(Hypothesis 1): Treatment-naïve women with Stage II-III breast cancer (without known brain metastases) will experience increased amount of neuroinflammation and greater cognitive decline after completing neodjuvant Chemotherapy Treatment (NACT).

(Hypothesis 2): Greater levels of neuroinflammation as measured by the amount and distribution of [18F]DPA-714 in the brain using PET/MRI after completing NACT will be associated with lower levels of cognitive functioning as measured by self-report and/or objective cognitive impairment/change.

Neuroinflammation will be measured using PET with tracer [18F]DPA-714 using a simultaneous PET/MRI system, and cognitive functioning will be measured with self-report and objective neuropsychological measures.

Exploratory Aim 2:

To investigate the relationships between CRCI and quality of life (QOL) and everyday functioning in breast cancer survivors after completing chemotherapy treatment.

For this Aim, we will assess QOL using self-report measures.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Female gender
3. Newly diagnosed treatment naïve women with stage II-III breast cancer that meet the following

   * Stage IIA: Any 1 of these conditions:

     * There is no evidence of a tumor in the breast, but the cancer has spread to 1 to 3 axillary lymph nodes. It has not spread to distant parts of the body. (T0, N1, M0)
     * The tumor is 20 mm or smaller and has spread to the axillary lymph nodes (T1, N1, M0)
     * The tumor is larger than 20 mm but not larger than 50 mm and has not spread to the axillary lymph nodes (T2, N0, M0)
   * Stage IIb: Either of these conditions

     * The tumor is larger than 20 mm but not larger than 50 mm and has spread to 1 to 3 axillary lymph nodes (T2, N1, M0)
     * The tumor is larger than 50 mm but has not spread to the axillary lymph nodes (T3, N0, M0)
   * Stage IIIA: The cancer of any size has spread to 4 to 9 axillary lymph nodes or to internal mammary lymph nodes. It has not spread to other parts of the body (T0, T1, T2, or T3, N2, M0. Stage IIIA may also be a tumor larger than 50 mm that has spread to 1 to 3 axillary lymph nodes (T3, N1, M0)
4. English is the primary language
5. Planned neoadjuvant chemotherapy that includes a taxane and/or an anthracycline drug as part of the treatment regimen.

Exclusion Criteria:

1. Contraindications to PET/MRI, including claustrophobia
2. Low-affinity binder for TSPO ligands when genotyping is available prior to PET imaging
3. Pregnancy
4. Lactation
5. Individuals who are unable to participate in the imaging portion due to the severity of their medical condition
6. Chronic infectious disease (e.g., HIV, HCV)
7. Chronic inflammatory disease (e.g., fibromyalgia, MS, etc) or autoimmune disease
8. Viral or bacterial illness requiring medical attention and/or antibiotics within 1 month of study participation
9. Blood or blood clotting disorder
10. Cancer that has metastasized to the brain
11. Positive urine β-hCG test day of the procedure or a serum-hCG test within 48 hours prior to the administration of [18F]DPA-714
12. Currently enrolled in a clinical trial utilizing experimental therapies.
13. Prior brain tumor or other neurological condition known to affect cognition
14. A diagnosis of dementia unrelated to cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Measure regional brain TSPO levels using [F-18]DPA-714-PET before and after neoadjuvant chemotherapy | Pre-study visit through completion of neoadjuvant chemotherapy (NACT) (Usually around 12 weeks)
  Levels will be presented with mean and 95% CI in the Freesurfer regions of interest (ROI), including cerebellum, hippocampus, amygdala, three white matter regions (frontal, parietal, and occipital), and three cortical gray matter regions (frontal, parietal, and occipital), by combining the corresponding sub-regions provided by Freesurfer.